CLINICAL TRIAL: NCT05354804
Title: Aiming Towards Evidence Based Interpretation of Cardiac Biomarkers in Patients Presenting With Chest Pain Using Point of Care Assays
Acronym: WESTCOR-POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 285544
Record Dates: First submitted 2022-03-22; First posted 2022-04-29 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2023-08

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Placebo Comparator): Patients randomized to standard care will be sampled at admission and after 1 hour (and furthermore as clinically indicated). High sensitive Troponin T (cTnT) and standard laboratory tests will be measured in the central hospital laboratory using Cobas e801 from Roche Diagnostics and eligibility for rule-out will be judged in accordance with the ESC 0/1 hour rule-out algorithm for cTnT. ECG and HEART-score will be obtained in all patients, other clinical investigations will be ordered by the attending physician. If NSTE-ACS is low risk based on the cTnT algorithm, HEART< 4 and non-ischemic ECG, patients will be investigated according to the ED flow chart for non-coronary acute chest pain, in order to identify differential diagnoses. Patients will be admitted or discharged based on the clinical judgement of the attending physician.
  Interventions: Diagnostic Test: Troponin T (Roche Diagnostics) 0/1 hour ESC algorithm
- POC (Active Comparator): Blood samples will be obtained at admission, standard blood tests will be measured at the central laboratory whilst high sensitive troponin I at 0 and 1 hour will be analyzed using a POC instrument from Siemens Healthineers in the ED. ECG and HEART-score will be obtained in all patients, other clinical investigations will be ordered by the attending physician. If the cTnI concentration at admission and the 1-hour delta is below a pre-specified concentration, the HEART- score < 4, and the ECG is non-ischemic the patients will be allocated to the rule-out of NSTEMI group and investigated according to the ED flow chart for non-coronary acute chest pain, in order to identify differential diagnosis. Finally, patients will be admitted or discharged based on the clinical judgement of the attending physician.
  Interventions: Diagnostic Test: Troponin I (Siemens VTli) 0/1 hour algorithm

INTERVENTIONS:
Diagnostic Test: Troponin I (Siemens VTli) 0/1 hour algorithm — Patients will be investigated using the ESC 0/1 hour cTnT algorithm from ESC compared to a 0/1 hour algorithm utilizing the Siemens VTli POC instrument for cTnI.
  Arms: POC
Diagnostic Test: Troponin T (Roche Diagnostics) 0/1 hour ESC algorithm — Patients will be investigated using the ESC 0/1 hour cTnT algorithm from ESC compared to a 0/1 hour algorithm utilizing the Siemens VTli POC instrument for cTnI.
  Arms: Standard

SUMMARY:
The aim of the current study is to perform a RCT comparing safety and efficiency of a standard care (in-line with current ESC recommendations) to an algorithm that utilize a POC troponin tests for bedside measurement, the instruments could be located in the ED and return results in few minutes.

DETAILED DESCRIPTION:
Ischemic coronary artery disease is an important health challenge and a common cause of death worldwide. Patients with symptoms suggestive of acute coronary syndrome are frequently referred to the emergency department (ED) and impose a high work-load on hospitals. Since 2009, high-sensitivity cardiac troponin (hs-cTn) assays have become a crucial ED tool for differentiating between patients with and without Non-ST-elevation myocardial infarction (NSTEMI). Accordingly, the European Society of Cardiology (ESC) recommends 0-1 hour algorithms that use hs-cTn for rule-out and rule-in of NSTEMI.

Additionally, the clinical suspicion of acute coronary syndrome (ACS) or other life-threating conditions must be low.

Unfortunately, these algorithms have been difficult to implement into routine and clinical practice, and are only used by a limited number of hospitals due to lack of randomized clinical trials and practical obstacles, including turnaround time for troponins.

The aim of the current study is to perform a RCT comparing safety and efficiency of a standard care (in-line with current ESC recommendations) to an algorithm that utilize a POC troponin tests for bedside measurement, the instruments could be located in the ED and return results in few minutes.

ELIGIBILITY:
Inclusion Criteria:

Patients > 17 years who are referred to the Emergency Department of Haukeland University Hospital with chest pain suspect of ACS

Exclusion Criteria:

1. STEMI (ECG criteria)
2. Patients without STEMI who are immediately transferred to cardiac catheterisation lab (due to heart failure, arrhythmia etc.) without possibility for blood sampling
3. Patients admitted from Nursing homes
4. Patients transferred from other hospitals (e.g. for PCI treatment)
5. Less than 2 months life expectancy from comorbid clinical conditions
6. Not possible to provide informed consent due to cognitive impairment, language problems or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1496 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Length of stay in the Emergency Department (ED) | Up to 24 hours
  Difference in length of stay in the ED will be compared between the two arms

SECONDARY OUTCOMES:
Discharge rate at 3 hours | 3 hours
  Percentages of patients who are discharged within 3 hours will be compared between the two arms
Discharge rate at 6 hours | 6 hours
  Percentages of patients who are discharged within 6 hours will be compared between the two arms
Total length of stay | Up to 3 months
  Time from arrival in the ED to discharge from hospital (hours) will be compared between the two arms
Composite of myocardial infarction and death | 30 days
  Differences in composite of death, myocardial infarction and acute revascularization within 30 days will be compared between the two arms.
Composite of myocardial infarction, death and revascularization | 30 days
  Death, myocardial infarction or acute revascularization within 12 months after inclusion will be compared between the two arms
Composite of myocardial infarction and death | 1 year
  Differences in composite of death, myocardial infarction and acute revascularization within 30 days will be compared between the two arms.
Composite of myocardial infarction, death and revascularization | 1 year
  Death, myocardial infarction or acute revascularization within 12 months after inclusion will be compared between the two arms
Total patient episode costs | Up to 3 months
  Total patient episode costs will be calculated and compared between the two arms
12 months costs | 12 months
  Costs related to all hospital contacts during 12 months follow-up
Patients quality of life according to RAND-12 | 30 days
  Patients quality of life will be measured 30 days after discharge using RAND-12 questionnaire and compared between the two arms.
Symptom burden | 30 days
  Patients quality of life will be measured 30 days after discharge using SAQ7 questionnaire and compared between the two arms
Patient satisfaction | 30 days
  Change in patients satisfaction with the hospital admission/contact will be measured 30 days after discharge using PasOP14 questionnaire and compared between the two arms

OTHER OUTCOMES:
Re-admission | 30 days
  Readmission of any cause within 30 days after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M Aakre, MD/PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data.